## Official Title: The Effect of EMG Activity on Anesthetic Depth Monitoring: Comparison Between Phase Lag Entropy and BIS

Date of the document: September 8th, 2017

NCT03230929

## Statistical Analysis Plan

Paired t-test could be used for verifying the statistical difference of the bispectral index (BIS) values and phase lag entropy (PLE) before and after sugammadex administration for reversal of muscle relaxation. We will proceed with the post-hoc test for BIS values and PLE measured at every 1 minute for 5 minutes after administration of sugammadex. If the P value is less than 0.05, it is interpreted as statistical significance.